CLINICAL TRIAL: NCT01815684
Title: A Phase I, Double Blind, Placebo-controlled, Randomized 4-way Alternating Cross-over Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of Single Ascending Doses of ASP3652 in Healthy Young Caucasian Male and Female Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Effects of Single Ascending Doses of ASP3652 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 3652-CL-0049; 2011-004247-41 (EudraCT Number)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Pharmacokinetics; Pharmacodynamics; Healthy Subjects; Safety
Keywords: Phase I; ASP3652; Dose escalation; Maximum Tolerated Dose (MTD)
MeSH Terms: interventions — ASP3652

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP3652 Group 1 (Experimental): Dosed according to the following scheme: placebo, low dose, medium dose, high dose
  Interventions: Drug: ASP3652; Drug: Placebo
- ASP3652 Group 2 (Experimental): Dosed according to the following scheme: low dose, placebo, medium dose, high dose
  Interventions: Drug: ASP3652; Drug: Placebo
- ASP3652 Group 3 (Experimental): Dosed according to the following scheme: low dose, medium dose, placebo, high dose
  Interventions: Drug: ASP3652; Drug: Placebo
- ASP3652 Group 4 (Experimental): Dosed according to the following scheme: low dose, medium dose, high dose, placebo
  Interventions: Drug: ASP3652; Drug: Placebo

INTERVENTIONS:
Drug: ASP3652 — Oral
Drug: Placebo — Oral

SUMMARY:
The purpose of this study is to explore the safety (including the effect on cardiac intervals), tolerability, the effects on the Central Nervous System (CNS), as well as the CNS side effect profile of single ascending doses of ASP3652 in healthy, Caucasian male and female subjects.

DETAILED DESCRIPTION:
Each subject receives 3 single ascending doses of ASP3652 and a single dose of matching placebo during one randomly selected investigational period. Randomization is conducted separately for males and females.

The washout period between dosing occasions is at least 7 days. Screening takes place from Day -22 to Day -2. Subjects are admitted to the clinic in the afternoon of Day -1 of investigational period 1, 2, 3 and 4 for pre-dose assessments.

On Day -1 of all investigational periods, subjects do not take any food or drink for at least 10 hours before the anticipated dosing time on Day 1. For the duration of their stay in the clinic, subjects are not allowed to consume caffeine or other xanthine-containing drinks.

The subjects are discharged on Day 4 of each investigational period. The End of Study Visit (ESV) is planned to take place 7-14 days after early discharge or after Day 4 of investigational period 4.

ELIGIBILITY:
Inclusion Criteria:

* Subject is white and of Caucasian origin.
* Body Mass Index more than or equal to 18.5 and less than 30.0kg/m2.
* Male subject must agree to practice an adequate contraceptive method with female sexual partners to prevent pregnancy.
* Female subject must agree to practice an adequate contraceptive method with male sexual partners to prevent pregnancy.

Exclusion Criteria:

* Pregnancy within 6 months before screening assessment or breast feeding within 3 months before screening (for females subjects only).
* Known or suspected hypersensitivity to ASP3652, or any components of the formulation used.
* A mean QTc(F) interval of >430 ms (for males) and >450 ms (for females) after triplicate measurements, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS). In case of an abnormal QTc(F) interval, the assessment may be repeated once (in triplicate). If the QTc(F) interval exceeds the limits, two additional Electrocardiogram (ECG)s can be recorded and the average of the three QTc(F) values should be used to determine the subject's eligibility.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses of ASP3652 assessed through vital signs, adverse events, electrocardiogram and clinical laboratory assessments | Day -22 to ESV (7-14 days after (early) discharge)
Safety and tolerability of single ascending doses of ASP3652 assessed through electrocardiogram | Day -22 to ESV (7-14 days after (early) discharge)
  QT (Q wave to T wave)/QTc interval (QT interval corrected for heart rate), QT interval, RR (R wave to R wave) interval, HR (Heart Rate), PR interval, QRS interval, QTcB, QTcF

SECONDARY OUTCOMES:
Pharmacokinetic profile of single ascending doses of ASP3652 | Days 1- 4 (Investigational period 1 - 4)
  Plasma: Cmax (Maximum concentration), AUClast (AUC until last sample taken), AUCinf (AUC extrapolated until infinity), tmax (Time to attain Cmax), tlag (Absorption lag time), t1/2 (Apparent terminal elimination half-life), Vz/F (Apparent volume of distribution), CL/F (Apparent total body plasma clearance)/ Urine: Aelast (Amount excreted in urine until last sample), Aeinf (Cumulative amount of unchanged drug excreted into the urine from time zero to infinity after single dose), Aelast% (Percentage of unchanged drug excreted into the urine from time of last measurable concentration), Aeinf% (Percentage of unchanged drug excreted into the urine from time zero to infinity after single dose), CLR (Renal clearance)
Effect of single ascending doses of ASP3652 on CNS Pharmacodynamics | Days 1 - 4 (Investigational period 1 - 4)
  Body sway, alertness, perception, mood, learning, memory, distraction, adaptive tracking, eye movements, addiction, neuro-endocrine parameters
Effect of single ascending doses of ASP3652 on plasma levels of enzyme substrates | Days 1 - 4 (Investigational period 1 - 4)
  Rmax, tmax R, AUR

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Takizawa M, Cerneus D, Michon I, Rijnders S, Meijer J, Someya A, Sato Y. Investigation of Safety and Tolerability of ASP3652 Based on Clinical Studies of Cerebrospinal Fluid Transfer After Multiple Doses and Exposure After Single Doses at High Dose Levels. Adv Ther. 2020 Sep;37(9):3967-3984. doi: 10.1007/s12325-020-01451-6. Epub 2020 Jul 26. PMID 32715381